CLINICAL TRIAL: NCT05508334
Title: An Open-label, Non-randomised, Multicentre Study to Allow Continued Access to and Assess the Safety and Tolerability of RC88 for Patients With Advanced Solid Tumours
Brief Title: A Study to Assess the Safety and Tolerability of RC88 for Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC88 C002
Record Dates: First submitted 2022-08-01; First posted 2022-08-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: RC88 (Experimental): Subjects will receive intravenous infusion of RC88 once every 2 weeks in a dose escalation fashion until confirmed progression, unacceptable toxicity, or any criterion for withdrawal from the trial or investigational medicinal product (IMP) occurs
  Interventions: Drug: RC88

INTERVENTIONS:
Drug: RC88 — Every 2 weeks for a maximum of 2 years
  Other Names: The injectable RC88

SUMMARY:
The purpose of this study is to allow RC88 treatment of patients with advanced solid tumours to assess the safety and tolerability of clinical pharmacology studies

DETAILED DESCRIPTION:
The main purpose of this Phase I study is to test RC88 at different dose levels to see if it is safe and well tolerated when given once every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must be ≥ 18 years at the first screening examination / visit.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
3. Life expectancy of at least 12 weeks
4. Phase I must be histologically or cytologically confirmed and have failed standard therapy (disease progression after treatment) or are intolerant,unable to receive, or nonexistent to standard care,Patients with partial,advanced or metastatic malignant solid tumors;
5. Phase II-Advanced malignant solid tumor with MSLN expression
6. Patients with malignant pleural mesothelioma were assessed using mRECIST criteria, and those with other cancers were assessed using RECIST V1.1 criteria
7. Phase II-Mesothelin (MSLN) positive as confirmed by the central laboratory.
8. Adequate organ function
9. Voluntarily sign an informed consent form

Exclusion Criteria:

1. Cancer metastases in the brain
2. Active infection or past hepatitis B or C infection
3. Major surgery less than 1 month before the start of the study
4. Uncontrolled heart disease
5. History of allergy to mesothelin-directed antibodies, tubulysin, monoclonal antibodies related compounds

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
RP2D | 28 days after first treatment
  Incidence of DLT (dose limiting toxicity) of RC88

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Maximum Concentration (Cmax) of RC88 | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 24, 48, 96, 168 hours
  Dose Escalation and Expansion Part
Terminal Half Life (t1/2) of RC88 | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 24, 48, 96, 168 hours
  Dose Escalation and Expansion Part
Progression Free Survival (PFS) | 24 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Remegen, Beijing, Beijing Municipality
  - Remgenen, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No